CLINICAL TRIAL: NCT00488787
Title: A Randomized, Double-Blind, Placebo-Controlled Pilot Study of the Safety and Efficacy of 10 mg, 30 mg, and 50 mg of Transnasal Ketamine Hydrochloride (PMI-100) for the Treatment of Postoperative Dental Pain
Brief Title: Safety and Efficacy of Intranasal Ketamine for the Treatment of Postoperative Dental Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Javelin Pharmaceuticals (Industry)
Responsible Party: Javelin Pharmaceuticals, Javelin Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KET-003
Record Dates: First submitted 2007-06-19; First posted 2007-06-20 (Estimated); Last update posted 2008-02-07 (Estimated); Status verified 2008-02

CONDITIONS: Pain, Postoperative
Keywords: dental; surgery; analgesia; 2-4 impacted third molars
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A (Experimental): Intranasal ketamine low dose
  Interventions: Drug: intranasal ketamine
- B (Experimental): intranasal ketamine medium dose
  Interventions: Drug: intranasal ketamine
- C (Experimental): intranasal ketamine high dose
  Interventions: Drug: intranasal ketamine
- D (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: intranasal ketamine — low dose
  Arms: A
Drug: intranasal ketamine — medium dose
  Arms: B
Drug: intranasal ketamine — high dose
  Arms: C
Drug: placebo — placebo
  Arms: D

SUMMARY:
Once patients' postoperative pain intensity reaches a moderate-to-severe level, they are randomized to receive intranasal ketamine or placebo. Patients remain in the study unit for 3 hours post administration and assess pain intensity and pain relief throughout the 3 hour postoperative period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients at least 16 years of age requiring two or more third molar extractions

Exclusion Criteria:

* Less than 16 years old
* Other exclusion criteria may apply

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2001-03; Primary Completion 2001-04 (Actual); Study Completion 2001-04 (Actual)

PRIMARY OUTCOMES:
total pain relief over 0-3 hours following dosing | 3 hours

SECONDARY OUTCOMES:
other pain assessments | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Christensen, DDS, Principal Investigator — Jean Brown Associates